CLINICAL TRIAL: NCT03007290
Title: Clinical Usefulness of Therapeutic Drug Monitoring of Colistin in Patients Treated With Colistin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eu Suk Kim, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Colistin_TDM
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Multidrug-resistant Gram-negative Bacteria Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Group with therapeutic drug monitoring
  Interventions: Other: Therapeutic drug monitoring

INTERVENTIONS:
Other: Therapeutic drug monitoring — Therapeutic drug monitoring for colistin

SUMMARY:
Clinical usefulness of therapeutic drug monitoring of colistin in patients treated with colistin

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Those who receive colistin therapy for the treatment of multi-drug resistant gram negative bacteria infection.

Exclusion Criteria:

* Those who received colistin therapy less than 48 hours
* Those who received colistin therapy through the bronchus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
AKI | Through study completion, an average of 1 month
  Emergence rate of acute kidney injury

SECONDARY OUTCOMES:
Death | Through study completion, an average of 1 month
  Death rate
Negative conversion rate | Through study completion, an average of 1 month
  Culture-negative conversion rate Treatment success Treatment success

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No